CLINICAL TRIAL: NCT04529278
Title: Efficacy and Tolerance of Liraglutide for Weight Loss in Obese Type 2 Diabetic Hemodialysis Patients
Acronym: LIRADIAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIRADIAL
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Hemodialysis; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liraglutide (Experimental): Liraglutide is initiated at 0.6 mg / day during week S1 (initiation D1) during weekly hospitalization in the diabetology department. Then the dose of liraglutide is increased to 1.2 mg / day on week S2 (increase in dose on D8) then to 1.8 mg / day on week S3 (increase in dose on D15).
  The daily dose is then 1.8 mg until week W26.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide is initiated at 0.6 mg / day during week S1 (initiation D1) during weekly hospitalization in the diabetology department. Then the dose of liraglutide is increased to 1.2 mg / day on week S2 (increase in dose on D8) then to 1.8 mg / day on week S3 (increase in dose on D15).
  The daily dose is then 1.8 mg until week W26.

SUMMARY:
Diabetes is the second leading cause of end stage renal disease in France (22% in the 2016 REIN register). In hemodialysis, its prevalence is higher, between 30-40% depending on the study. Associated with type 2 diabetes, a large number of patients present with overweight (body mass index or BMI> 25 kg / m2) which can lead to a temporary contraindication to kidney transplant by the surgeon, or even definitive once BMI is over 30 kg / m2. Indeed, above this threshold, patients are exposed to an increased risk of surgical complications (wall infections, suture release), hospitalizations and potentially transplant failure. A recent study based on the Kidney Registry showed that patients with a BMI> 31 kg / m2 were more likely to stay on dialysis than to benefit from a transplant whereas for each decrease of 1 kg / m2 of BMI, there is a 9-11% increase in the likelihood of being transplanted. The management of obesity in dialysis patients is important for reducing cardiovascular risks but also because it increases the chances of access to transplantation. However, current weight loss programs are disappointing. The changes in hygiene and diet rules integrated into a specialized monitoring program only allow a weight loss of 2 to 8% in 24 months for half of the patients. Bariatric surgery is, of course, a more effective alternative, but with a 10% risk of postoperative complications.

Glucagon-Like Peptide 1 (aGLP1) analogues are a new class of antidiabetic drugs that have revolutionized the management of type 2 diabetes. In fact, they combine efficacy on glycemic control but also on weight loss. They are used in obese non-diabetic people in some countries, with a reduction in weight of up to 10 to 15% with certain molecules. In addition, they have shown an effect on reducing cardiovascular events in diabetics including with Chronic Kidney Disease CKD 3-4. AGPL1 are well tolerated with side effects mainly of digestive tropism such as nausea or vomiting. Exceptionally, these effects can occur from the first injection requiring permanent discontinuation of treatment. In 20% of cases, these side effects can appear in the first weeks. They gradually fade, spontaneously or after symptomatic treatment and allow titration of the drug.

AGLP1 is currently contraindicated in patients with reduced renal function, that is, when the glomerular filtration rate (GFR) is <15 ml / min (MRC stage 5-5D), because this population specific was excluded from the originator studies. However, aGLP1 are small peptides that are not eliminated by the kidneys. Their elimination takes place through the general catabolism of proteins. To date, 2 publications have evaluated the safety profile and efficacy of an aGLP1, liraglutide (Victoza®), in diabetic dialysis patients. These studies showed that the 24 hour plasma concentration of liraglutide increased by 50% over the long term. The safety profile was acceptable with, as expected, a predominance of gastrointestinal effects in the first weeks of treatment such as nausea, vomiting. The authors suggest an adjustment of the dosages and a longer titration period to limit side effects. However, treatment with aGPL1 is effective with better glycemic control and an average weight loss of 2.6 kg over a period of 3 months. Studies show that weight loss under liraglutide continues beyond 3 months with possible losses between 4 and 8 kg at 6 months and 12 months of treatment followed 12. Liraglutide (Victoza®) is the analogue of GPL1 for which we have a sufficiently long follow-up (> 10 years) on its effectiveness and its short and long-term side effects.

The main objective of this project, in type 2 diabetic patients on dialysis, as a temporary contraindication for transplant due to overweight, is on the one hand to study the effect of liraglutide on weight loss and control of diabetes, and on the other hand to assess its tolerance in this population. The expected benefit is to be able to facilitate registration on the waiting list and access to renal transplantation of these overweight patients, without having to resort to more invasive methods such as bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 and <70
* Patient on hemodialysis for more than 6 months
* Type 2 diabetic patient
* Patient with a BMI> 30 kg / m2 with a Temporary Contraindication for kidney transplant for renal transplant due to overweight by his graft center
* Patient affiliated to a health insurance plan
* French speaking patient
* Patient having given free, informed and written consent

Exclusion Criteria:

* Patient with a Temporary Contraindication for kidney transplant for a cause other than overweight
* Patient with personal or family history of thyroid medullary cancer
* Patient with a history of acute or chronic pancreatitis
* Patient who has already had hypersensitivity to liraglutide (or to any other component of the product)
* Patient who has already had a severe digestive intolerance to taking GLP-1 receptor agonists (such as exenatide or lixisenatide)
* Patient already included in an interventional risk research protocol (RIPH1)
* Pregnant or lactating woman
* Patient under guardianship or curatorship
* Patient deprived of liberty

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight Loss at Week 26 | Week 26
  This outcome corresponds to Assess weight loss in obese diabetic patients on hemodialysis after 6 months of treatment with liraglutide in order to facilitate access to renal transplants for patients who have been rejected for being overweight.

SECONDARY OUTCOMES:
Lift of CIT for transplant for obesity | Week 26
  This outcome corresponds to establish the number and percentage of patients whose CIT transplant for obesity will be lifted after 6 months of treatment.
Tolerance of luraglutide | Week 26
  This outcome corresponds to evaluate the number and percentage of serious and non-serious adverse events in type 2 diabetic patients on hemodialysis.
Regulation of blood sugar | Week 26
  This ouctome correspond to evaluate the reducing the number / dose of anti-diabetic drugs or the daily dose of insulin.
Glycemic balance | Week 26
  This ouctome correspond to compare the average variations in glycated hemoglobin (HbA1c) between M0 and M6.
Hypoglycemia | Week 26
  This ouctome correspond to evaluate the percentage of hypoglycaemia between Week 1 and Week 26.
Evolution of weight | Week 26
  This ouctome corresponds to evaluate the modifications of the dry mass and the fatty mass between M0 and M6 by bioimpedancemetry.
Therapeutic monitoring | Week 26
  This ouctome corresponds to evaluateconcentration of liraglutide before and after the dialysis session.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Touzot, MD, Study Director — AURA Paris Plaisance
Locations (4):
- France (4):
  - AURA Paris Plaisance, Paris, Groupe Hospitalier Paris Saint-Joseph
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Hôpital Bichat, Paris
  - AURA Paris Site de Saint Ouen, Saint-Ouen

REFERENCES:
- [Result] Nicoletto BB, Fonseca NK, Manfro RC, Goncalves LF, Leitao CB, Souza GC. Effects of obesity on kidney transplantation outcomes: a systematic review and meta-analysis. Transplantation. 2014 Jul 27;98(2):167-76. doi: 10.1097/TP.0000000000000028. PMID 24911038
- [Result] Gill JS, Hendren E, Dong J, Johnston O, Gill J. Differential association of body mass index with access to kidney transplantation in men and women. Clin J Am Soc Nephrol. 2014 May;9(5):951-9. doi: 10.2215/CJN.08310813. Epub 2014 Apr 17. PMID 24742478
- [Result] Lassalle M, Fezeu LK, Couchoud C, Hannedouche T, Massy ZA, Czernichow S. Obesity and access to kidney transplantation in patients starting dialysis: A prospective cohort study. PLoS One. 2017 May 11;12(5):e0176616. doi: 10.1371/journal.pone.0176616. eCollection 2017. PMID 28493926
- [Result] MacLaughlin HL, Cook SA, Kariyawasam D, Roseke M, van Niekerk M, Macdougall IC. Nonrandomized trial of weight loss with orlistat, nutrition education, diet, and exercise in obese patients with CKD: 2-year follow-up. Am J Kidney Dis. 2010 Jan;55(1):69-76. doi: 10.1053/j.ajkd.2009.09.011. Epub 2009 Nov 17. PMID 19926371
- [Result] Turgeon NA, Perez S, Mondestin M, Davis SS, Lin E, Tata S, Kirk AD, Larsen CP, Pearson TC, Sweeney JF. The impact of renal function on outcomes of bariatric surgery. J Am Soc Nephrol. 2012 May;23(5):885-94. doi: 10.1681/ASN.2011050476. Epub 2012 Mar 1. PMID 22383694
- [Result] Nauck M, Frid A, Hermansen K, Shah NS, Tankova T, Mitha IH, Zdravkovic M, During M, Matthews DR; LEAD-2 Study Group. Efficacy and safety comparison of liraglutide, glimepiride, and placebo, all in combination with metformin, in type 2 diabetes: the LEAD (liraglutide effect and action in diabetes)-2 study. Diabetes Care. 2009 Jan;32(1):84-90. doi: 10.2337/dc08-1355. Epub 2008 Oct 17. PMID 18931095
- [Result] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305
- [Result] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Result] Mann JFE, Orsted DD, Brown-Frandsen K, Marso SP, Poulter NR, Rasmussen S, Tornoe K, Zinman B, Buse JB; LEADER Steering Committee and Investigators. Liraglutide and Renal Outcomes in Type 2 Diabetes. N Engl J Med. 2017 Aug 31;377(9):839-848. doi: 10.1056/NEJMoa1616011. PMID 28854085
- [Result] Idorn T, Knop FK, Jorgensen MB, Jensen T, Resuli M, Hansen PM, Christensen KB, Holst JJ, Hornum M, Feldt-Rasmussen B. Safety and Efficacy of Liraglutide in Patients With Type 2 Diabetes and End-Stage Renal Disease: An Investigator-Initiated, Placebo-Controlled, Double-Blind, Parallel-Group, Randomized Trial. Diabetes Care. 2016 Feb;39(2):206-13. doi: 10.2337/dc15-1025. Epub 2015 Aug 17. PMID 26283739
- [Result] Osonoi T, Saito M, Tamasawa A, Ishida H, Tsujino D, Nishimura R, Utsunomiya K. Effect of hemodialysis on plasma glucose profile and plasma level of liraglutide in patients with type 2 diabetes mellitus and end-stage renal disease: a pilot study. PLoS One. 2014 Dec 19;9(12):e113468. doi: 10.1371/journal.pone.0113468. eCollection 2014. PMID 25526642
- [Result] Overbeek JA, Heintjes EM, Huisman EL, Tikkanen CK, van Diermen AW, Penning-van Beest FJA, Herings RMC. Clinical effectiveness of liraglutide vs basal insulin in a real-world setting: Evidence of improved glycaemic and weight control in obese people with type 2 diabetes. Diabetes Obes Metab. 2018 Sep;20(9):2093-2102. doi: 10.1111/dom.13335. Epub 2018 May 29. PMID 29726082